CLINICAL TRIAL: NCT06446440
Title: Comperative Study Between Laparoscopic Adhesiolysis Vs Open Adhesiolysis in Adhesive Intestinal Obstruction
Brief Title: Lap Adhesiolysis in Intestinal Obstruction
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Bemen Soliman Haroun Abdulla, General Surgery department at assiut University hospitals, Assiut University
Other Study IDs: Lap adhesiolysis
Record Dates: First submitted 2024-06-01; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Adhesions Bowel

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: These group will include cases underwent laparoscopic adhesiolysis
  Interventions: Procedure: Laparoscopic adhesiolysis
- Group B: These group will include cases underwent open adhesiolysis
  Interventions: Procedure: Open adhesiolysis

INTERVENTIONS:
Procedure: Laparoscopic adhesiolysis — Laparoscopic adhesiolysis
  Groups: Group A
Procedure: Open adhesiolysis — Open adhesiolysis
  Groups: Group B

SUMMARY:
Comparison between the results of laparotomy and laparoscopy in adhesive intestinal obstruction and introduce the use of laparoscopy to the emergency setting in Asyut University Hospital.

DETAILED DESCRIPTION:
Adhesive Intestinal obstruction is one of the most common complications after any abdominal surgery.

Adhesions account for 75% of causes of intestinal obstruction. laparoscopic adhesiolysis recently increase in frequency over open adhesiolysis but there is no definit evidence of its superiority. In term of length of hospital stay and morbidity.

adhesive bowel obstruction mainly managed by conservative treatment but some refractory cases needs surgical intervention In this study we will evaluate feasibility and efficacy of using laparoscop in adhesiolysis over open approach .

ELIGIBILITY:
Inclusion Criteria:

* any male or female above 18 years has adhesive Intestinal obstruction
* patient fulfilled the criteria to participate but operated before time of study if adequate data available
* patient in which conservative management is failed

Exclusion Criteria:

* othe casues of intestinal obstruction (other than adhsions)
* shocked patient
* cardiovascular diseases
* coagulopathy
* liver cirrhosis
* intracranial diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any case of intestinal obstruction and failed medical treatment and for surgery either open or laparoscopic adhesiolysis
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | 2 years
  Signs and symptoms of intestinal obstruction

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided